CLINICAL TRIAL: NCT02721069
Title: A 12-Month Open-Label, Repeat-Dose Safety Study of NRL-1 in Epilepsy Subjects (DIAZ.001.05)
Brief Title: Repeat Dose Safety Study of NRL-1 in Epilepsy Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Neurelis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIAZ.001.05
Record Dates: First submitted 2016-03-17; First posted 2016-03-28 (Estimated); Results first posted 2022-01-31 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Acute Repetitive Seizures; Breakthrough Seizures
Keywords: Seizures; Epilepsy
MeSH Terms: conditions — Seizures; Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NRL-1 (Experimental): Intranasal dose of NRL-1 will be administered at either 5 mg, 10 mg, 15 mg, or 20 mg based on the subject's body weight.
  Interventions: Drug: NRL-1

INTERVENTIONS:
Drug: NRL-1
  Other Names: Intranasal diazepam

SUMMARY:
This is a 12 month safety study to evaluate the safety of repeated doses of NRL-1

DETAILED DESCRIPTION:
This is a Phase 3, repeat dose, open-label, safety study in Epilepsy subjects who have frequent breakthrough seizures or Acute Repetitive Seizures (ARS). NRL-1 will be administered as needed to treat bouts of those seizures over a 12-month period of time. Doses will be defined as 5 mg, 10 mg, 15 mg, or 20 mg based on the subject's body weight. A diary will be used to record the seizure and NRL-1 administration.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects between the ages of 6 and 65 years, inclusive.
2. Written informed consent to participate in the study.
3. Subject has a clinical diagnosis of Epilepsy and while on a stable regimen of anti-epileptic medication, still experiences bouts of seizures (e.g. frequent break through seizures or Acute Repetitive Seizures [ARS]), and who, in the opinion of the Investigator, may need benzodiazepine intervention for seizure control at least 1 time a month on average.
4. Subject has a qualified caregiver or medical professional available that can administer study medication in the event of a seizure.
5. Subjects having either partial or generalized Epilepsy with motor seizures or seizures with clear alteration of awareness.
6. Female subjects of childbearing potential, defined as having a menstrual cycle and who are not surgically sterile or less than two (2) years postmenopausal, must complete a pregnancy screen and agree to utilize one of the following forms of contraception during the trial and for 21 days after the last dose of study drug: abstinence, hormonal (oral, transdermal, implant, or injection), barrier (condom, diaphragm with spermicide), intrauterine device (IUD), or vasectomized partner (six months minimum). Subjects must have used the same method for at least one (1) month prior to starting the study.
7. No clinically significant abnormal findings in the medical history, on the physical examination or electrocardiogram (QTcF<450 msec for males and QTcF<470 msec for females).
8. Subjects and caregivers must agree to return to the study site for all study visits and must be willing to comply with all required study procedures.

Exclusion Criteria:

1. A history of clinically significant gastrointestinal, renal, hepatic, hematologic, endocrine, oncologic, pulmonary, immunologic, psychiatric, or cardiovascular disease, or any other condition which, in the opinion of the Investigator, would jeopardize the safety of the subject.
2. Subject has had significant traumatic injury, major surgery or open biopsy within 30 days prior to study screening.
3. Subjects with active major depression or a past suicide attempt, or any Suicidal Ideation of 3, 4, or 5 or any Suicidal Behavior in Lifetime using Columbia-Suicide Severity Rating Scale (C-SSRS). The pediatric C-SSRS should be used for subjects age 6 to 11. The adult C SSRS should be used for subjects 12 and greater years of age.
4. A history of allergic or adverse responses to diazepam or any comparable or similar product.
5. Participation in a clinical trial other than protocol DIAZ.001.04 within 30 days prior to Day 0. Participation in an observational (non-interventional) study is not excluded as long as there are no scheduling conflicts with this study.
6. Positive serum pregnancy test (ß-hCG) at screening for subjects age 12 or greater.
7. Positive blood screen for Human immunodeficiency virus (HIV), Hepatitis B surface antigen (HbSAg), or Hepatitis C, or a positive urine screen for alcohol or drugs of abuse, except marijuana use for medical reasons. When marijuana was used for medical reasons in the opinion of the investigator, it is not considered as drug abuse and the patient can be enrolled even if the marijuana metabolites in the urine revealed as positive.

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2016-04-11 (Actual); Primary Completion 2020-06-17 (Actual); Study Completion 2020-07-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Clinical Trials, Inc., Little Rock, Arkansas
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - New York University Comprehensive Epilepsy Center, New York, New York
  - Thomas Jefferson University Hospital Laboratory, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Misra SN, Jarrar R, Stern JM, Becker DA, Carrazana E, Rabinowicz AL. Rapid Rescue Treatment with Diazepam Nasal Spray Leads to Faster Seizure Cluster Termination in Epilepsy: An Exploratory Post Hoc Cohort Analysis. Neurol Ther. 2024 Feb;13(1):221-231. doi: 10.1007/s40120-023-00568-4. Epub 2024 Jan 4. PMID 38175488
- [Derived] Tarquinio D, Wheless JW, Segal EB, Misra SN, Rabinowicz AL, Carrazana E. Safety of Diazepam Nasal Spray in Pediatric Patients With Developmental Epileptic Encephalopathies: Results From a Long-term Phase 3 Safety Study. J Child Neurol. 2023 May;38(6-7):389-393. doi: 10.1177/08830738231185424. Epub 2023 Jul 16. PMID 37455404
- [Derived] Cramer JA, Faught E, Davis C, Misra SN, Carrazana E, Rabinowicz AL. Quality-of-life results in adults with epilepsy using diazepam nasal spray for seizure clusters from a long-term, open-label safety study. Epilepsy Behav. 2022 Sep;134:108811. doi: 10.1016/j.yebeh.2022.108811. Epub 2022 Jul 8. PMID 35816831
- [Derived] Wheless JW, Miller I, Hogan RE, Dlugos D, Biton V, Cascino GD, Sperling MR, Liow K, Vazquez B, Segal EB, Tarquinio D, Mauney W, Desai J, Rabinowicz AL, Carrazana E; DIAZ.001.05 Study Group. Final results from a Phase 3, long-term, open-label, repeat-dose safety study of diazepam nasal spray for seizure clusters in patients with epilepsy. Epilepsia. 2021 Oct;62(10):2485-2495. doi: 10.1111/epi.17041. Epub 2021 Aug 21. PMID 34418086
- [Derived] Miller I, Wheless JW, Hogan RE, Dlugos D, Biton V, Cascino GD, Sperling MR, Liow K, Vazquez B, Segal EB, Tarquinio D, Mauney W, Desai J, Rabinowicz AL, Carrazana E; DIAZ.001.05 Study Group. Consistent safety and tolerability of Valtoco(R) (diazepam nasal spray) in relationship to usage frequency in patients with seizure clusters: Interim results from a phase 3, long-term, open-label, repeat-dose safety study. Epilepsia Open. 2021 Sep;6(3):504-512. doi: 10.1002/epi4.12494. Epub 2021 May 13. PMID 34033266
- [Derived] Penovich P, Wheless JW, Hogan RE, Guerra C, Cook DF, Carrazana E, Rabinowicz AL. Examining the patient and caregiver experience with diazepam nasal spray for seizure clusters: Results from an exit survey of a phase 3, open-label, repeat-dose safety study. Epilepsy Behav. 2021 Aug;121(Pt A):108013. doi: 10.1016/j.yebeh.2021.108013. Epub 2021 May 19. PMID 34022621

RESULTS

PARTICIPANT FLOW:
Groups:
- NRL-1: Intranasal dose of NRL-1 will be administered at either 5 mg, 10 mg, 15 mg, or 20 mg based on the subject's body weight.
  NRL-1
Period: Overall Study
Arm/Group | NRL-1
Started | 175
Completed | 117
Not Completed | 58

BASELINE CHARACTERISTICS:
Arm/Group | NRL-1
Number analyzed (Participants) | 175
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 92
  Between 18 and 65 years | 82
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.3 (14.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93
  Male | 82
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 5
  Black or African American | 19
  White | 143
  More than one race | 4
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 175

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Received NRL-1 (Valtoco)
Description: Assess the number of participants who received at least one dose of NRL-1 (Valtoco) during the study and comprised the safety population.
Time Frame: 12 months
Population: Subjects who received at least one dose of NRL-1.
Measure: Count of Participants; unit: Participants
Groups:
- NRL-1 5mg: Intranasal dose of NRL-1 will be administered at 5 mg based on age and weight.
- NRL-1 10mg: Intranasal dose of NRL-1 will be administered at 10 mg based on age and weight.
- NRL-1 15 mg: Intranasal dose of NRL-1 will be administered at 15 mg based on age and weight.
- NRL-1 20mg: Intranasal dose of NRL-1 will be administered at 20 mg based on age and weight.
Arm/Group | NRL-1 5mg | NRL-1 10mg | NRL-1 15 mg | NRL-1 20mg
Number analyzed (Participants) | 11 | 61 | 46 | 57
Participants | 9 | 54 | 46 | 54

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- NRL-1 5mg; NRL-1 10mg; NRL-1 15mg; NRL-1 20mg: Intranasal dose of NRL-1 will be administered at 5, 10, 15, and 20 mg based on age and weight.
Arm/Group | NRL-1 5mg | NRL-1 10mg | NRL-1 15mg | NRL-1 20mg
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/54 | 0/46 | 1/54
Serious Adverse Events (participants affected / at risk) | 2/9 | 20/54 | 15/46 | 13/54
Other Adverse Events (participants affected / at risk) | 6/9 | 34/54 | 24/46 | 21/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NRL-1 5mg (N=9) | NRL-1 10mg (N=54) | NRL-1 15mg (N=46) | NRL-1 20mg (N=54)
Seizure (Nervous system disorders) | 1 (1) | 11 (16) | 8 (14) | 4 (5)
Status Epilepticus (Nervous system disorders) | 0 (0) | 5 (7) | 1 (1) | 1 (2)
Epilepsy (Nervous system disorders) | 0 (0) | 2 (3) | 1 (2) | 2 (3)
Seizure Cluster (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disturbance in Attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lennox-Gastaut Syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle Spasticity (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Partial Seizures (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Petit Mal Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postictal State (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large Intestinal Ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint Dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thermal Burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wrist Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sudden Unexplained Death in Epilepsy (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Restrictive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colorectal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hallucination, Visual (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Major Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Feeding Disorder (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine Haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mitral Valve Prolapse (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Brain Lobectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 4 (4) | 1 (3) | 2 (2)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis Perforated (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colonic Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis Streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NRL-1 5mg (N=9) | NRL-1 10mg (N=54) | NRL-1 15mg (N=46) | NRL-1 20mg (N=54)
Nasopharyngitis (Infections and infestations) | 1 (3) | 12 (13) | 3 (3) | 4 (6)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 9 (10) | 7 (8) | 4 (4)
Influenza (Infections and infestations) | 3 (4) | 5 (5) | 3 (3) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (2) | 4 (8) | 3 (3) | 3 (4)
Seizure (Nervous system disorders) | 0 (0) | 4 (5) | 7 (8) | 2 (4)
Somnolence (Nervous system disorders) | 0 (0) | 5 (5) | 4 (4) | 2 (2)
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (11) | 6 (16)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 4 (4) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (5) | 2 (2) | 2 (4)
Pyrexia (General disorders) | 1 (1) | 10 (10) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-09-28): https://cdn.clinicaltrials.gov/large-docs/69/NCT02721069/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-08): https://cdn.clinicaltrials.gov/large-docs/69/NCT02721069/SAP_001.pdf